CLINICAL TRIAL: NCT02675166
Title: SALTO -2 ( Long Term Monitoring In Oncology ) : Getting Long-term Management of Adult Children Cured of Childhood Cancer in Rhône-Alpes, Multicentric Study
Brief Title: Getting Long-term Management of Adult Children Cured of Childhood Cancer in Rhône-Alpes
Acronym: SALTO-2
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1508056; 2015-A00656-43 (Other: ANSM)
Record Dates: First submitted 2016-01-22; First posted 2016-02-05 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Pediatric Cancer; Sequels; Complications
Keywords: Childhood cancer; Sequels; Complications; Surgery; Radiotherapy; Chemotherapy; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric cancer young adult survivors: 544 patients alive and that are min 18 years old, included in the ARCERRA population register, for a primary cancer (not leukemia), diagnosed between 15 years old, between January the 1st 1993, and December the 31st 1999, in Rhône-Alpes.
  Interventions: Other: Pediatric cancer young adult survivors

INTERVENTIONS:
Other: Pediatric cancer young adult survivors — Patients will receive a questionnaire, a consultation with an oncologist and a psychologist will be planned, and two years later, patients will have to answer again to the questionnaire.
  Other Names: Long term follow up

SUMMARY:
Children cancers are rare and survival rate are around 75%. 1 French adult out of 850 is estimated as a children-cancer-survivor. Chemotherapy, radiotherapy or surgical complications can lead to a late risk of death. A regularly support, a therapeutic education, a support of the psychological difficulties have a positive impact on the quality of life and on long-term health for patients surviving to a cancer.

The ARCERRA exists, registering around 150 new cases a year. They coordinated, from 2011 to 2014, a multicentric study with a long term follow up in oncology (SALTO). 150 patients diagnosed between 1987 and 1992 were included, and the study demonstrated the feasibility and utility for patients and their physicians of a long-term follow-up coupled with an interview with a psychologist in Rhône-Alpes-Auvergne.

The primary objective of SALTO-2 project is to know the becoming of young adults that survived to pediatric cancer, diagnosed in Rhône-Alpes between 1993 and 1999. The second objective is in one hand to study the psychological becoming and on another hand, to ameliorate their lifestyle thanks to different documents created specially for them.

DETAILED DESCRIPTION:
Children cancers are rare and survival rate are around 75%. 1 French adult out of 850 is considered as a children-cancer-survivor. Chemotherapy, radiotherapy or surgical complications can lead to a late risk of death estimated in literature at 14%. A regularly support, a therapeutic education, a support of the psychological difficulties have a positive impact on the quality of life and on long-term health for patients surviving to a cancer. Many countries developed structures able to take care for a long term this kind of patients. In France, such structures are going to be developed.

The register of cancers concerning children of Rhône-Alpes (ARCERRA) exists since 1987, registering around 150 new cases a year. They coordinated, from 2011 to 2014, a multicentric study with a long term follow up in oncology (SALTO). 150 patients diagnosed between 1987 and 1992 were included, and the study demonstrated the feasibility and utility for patients and their physicians of a long-term follow-up coupled with an interview with a psychologist in Rhône-Alpes-Auvergne.

The primary objective of SALTO-2 project is to know the becoming of young adults that survived to pediatric cancer, diagnosed in Rhône-Alpes between 1993 and 1999. The second objective is in one hand to study the psychological becoming and on another hand, to ameliorate their lifestyle thanks to different documents created specially for them.

This is a prospective cohort study of patients surviving cancer (excluding leukemia) diagnosed between 1993 and 1999 in the Rhône- Alpes region before age 15 years. A questionnaire concerning their general situation and their professional life, their shape, and their quality of life will be sent to them. A consultation with an oncologist and an internist if possible will be planned. The two physicians will adapt the consultation according to the SFCE (French society of struggle against cancers and leukemia of children and teenagers) recommendations. They will give the two SFCE's documents.

After that, a consultation with a psychologist will be proposed, with a questionnaire MINI evaluating psychological aspect.

Two years later, a new questionnaire will be delivered to the patients, to check the new events during this period. It will be added to a satisfaction survey, allowing the measure of documents' impact.

The results will allow the description of the long term impacts for these patients, to answer their eventually questions.

ELIGIBILITY:
Inclusion Criteria:

* Had a cancer diagnostic between January the 1st 1993 and December the 31st 1999, before the age of 15 years old, in Rhône-Alpes
* Being a beneficiary of health insurance
* Having signed the informed consent form

Exclusion Criteria:

* Having been diagnosed with leukemia as a primary cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is composed of 544 patients registered in the ARCERRA documùent. They survived at a pediatric cancer, diagnosed in Rhône-Alpes between January the 1st 1993 and December the 31st 1999. They were less than 15 years old during this period.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Medical complications (post cancer treatment) | 15 years after the end of the cancer treatment
  The investigators note the medical complications from the end of their cancer treatment to the inclusion visit. Theses complications depend on the type of treatment received.

SECONDARY OUTCOMES:
MINI questionnaire score | 15 years after the end of the cancer treatment
  The investigators measured the psychological complications (post cancer treatment) by MINI questionnaire score.
MINI questionnaire score | 17 years after the end of the cancer treatment
  The investigators measured the psychological complications (post cancer treatment) by MINI questionnaire score.
Quality of life : SF-36 scale | 15 years after the end of the cancer treatment
  Researchers will focus on the quality of life (measured with the SF-36 scale).
Quality of life : SF-36 scale | 17 years after the end of the cancer treatment
  Researchers will focus on the quality of life (measured with the SF-36 scale).

CONTACTS AND LOCATIONS:
Overall Officials: BERGER Claire, MD, Principal Investigator — CHU SAINT-ETIENNE; Léonie CASAGRANDA, PhD, Study Chair — CHU SAINT-ETIENNE
Locations (4):
- France (4):
  - Chu Grenoble, Grenoble
  - IHOP1 de Lyon, Lyon
  - CH Lyon Sud - Pierre Bénite, Lyon
  - Chu Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tardy F, Casagranda L, Protiere A, Buisson-Papet G, Garcin A, Trombert-Paviot B, Freycon C, Marec-Berard P, Massoubre C, Berger C. Long-Term Clinical and Psychiatric Complications of Young Adults Cured of a Pediatric Bone Tumor Diagnosed Between 1987 and 1999 in Rhone: Alpes Region (France). J Adolesc Young Adult Oncol. 2022 Dec;11(6):571-579. doi: 10.1089/jayao.2021.0145. Epub 2022 Jan 18. PMID 35049375